CLINICAL TRIAL: NCT05717569
Title: Stoss Therapy Versus Weekly Regimen of Vitamin D in Treatment of Children With Chronic Liver Disease
Brief Title: Different Regimens of Vitamin D in Treatment of Children With Chronic Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hebatallah Saad Mahmoud Ahmed, Assisstant lecturer of pediatrics ,Ain shams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: vitaminD in liver diseases
Record Dates: First submitted 2022-11-18; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Chronic Liver Disease and Cirrhosis
Keywords: vitamin D; fibroscan
MeSH Terms: conditions — Fibrosis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A: Stoss vitamin D therapy
  Interventions: Drug: Vitamin D
- Group B (Active Comparator): Group B: Oral vitamin D therapy .
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — o Fibroscan: as a non-invasive imaging study for measuring liver cirrhosis by transducer probe-induced elastic share wave that propagates through liver tissue to measure its velocity. It is a promising non-invasive method for detection of cirrhosis in patients with chronic liver disease. Therefore, fibroscan can be used regarding the decision of treatment and follow-up of patients with cirrhosis for screening and detection of the complications . In our study the investigators will assess liver fibrosis before and after vitamin D therapy using fibroscan.
  Other Names: Fibroscan

SUMMARY:
The primary aim is to assess the efficacy of two different Vitamin D regimes in the treatment of vitamin D deficiency in children with chronic liver disease. The secondary aim is to evaluate the effect of vitamin D on liver fibrosis utilizing fibroscan..

DETAILED DESCRIPTION:
• In this study, the investigators are going to find out the optimum regimen to be used for effective treatment of vitamin D deficiency in those patients and to study the effect of vitamin D treatment on liver fibrosis.

Vitamin D is a hormone involved in the regulation of mineral homeostasis. It protects skeletal integrity and modulates cell growth and differentiation . It is lipid soluble in nature and interacts with vitamin D receptors and regulates the expression of more than 200 genes, mostly involved in apoptosis, cell growth, and cell differentiation .

Fibroscan: as a non-invasive imaging study for measuring liver cirrhosis by transducer probe-induced elastic share wave that propagates through liver tissue to measure its velocity. It is a promising noninvasive method for detection of cirrhosis in patients with chronic liver disease. Therefore, fibroscan can be used regarding the decision of treatment and follow-up of patients with cirrhosis for screening and detection of the complications . In our study the investigators will assess liver fibrosis before and after vitamin D therapy using fibroscan.

Group A: who received stoss parenteral vitamin D therapy (200.000 IU) once followed by 600 IU/ day orally (equivalent to RDA as maintenance).

Group B: who received 50.000 IU/ week vitamin D orally for four weeks followed by the maintenance dose.

The total duration of therapy was 6 months in both groups .

ELIGIBILITY:
Inclusion Criteria:

Children below the age of 18 with chronic liver disease.

Exclusion Criteria:

* Patients with concomitant renal affection.
* Patients who are on anticonvulsant therapy.
* Patients who lost follow up
* Patients refuse to participate at any time throughout the study period.
* Non-compliant patients for more than 50% of time.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Vitamin D3 level after each regimen | six months
  Quantitative estimation of 25(OH)D level was done using enzyme-linked immunoassay (ELISA) before and after therapy will be done.

SECONDARY OUTCOMES:
Assessment of liver fibrosis by fibroscan | six months
  Fibroscan will be done for both groups before and after vitamin D therapy to assess the degree of fibrosis by using probes according to the patient's chest diameter and plotting the results on kilo pascal with the Metavir score. Thus assessment of the effect of vitamin D by both regimes on halting the progression of liver fibrosis if found.

CONTACTS AND LOCATIONS:
Overall Officials: Tawhida Abdel-Ghaffar, Professor, Study Chair — Ain Shams University
Locations (2):
- Egypt (2):
  - Ain shams university, Cairo
  - EL Demerdash Hospital ,Ain Shams university, Cairo

REFERENCES:
- [Background] Ratziu V, Bellentani S, Cortez-Pinto H, Day C, Marchesini G. A position statement on NAFLD/NASH based on the EASL 2009 special conference. J Hepatol. 2010 Aug;53(2):372-84. doi: 10.1016/j.jhep.2010.04.008. Epub 2010 May 7. No abstract available. PMID 20494470
- [Background] Gonzalez-Padilla E, Soria Lopez A, Gonzalez-Rodriguez E, Garcia-Santana S, Mirallave-Pescador A, Groba Marco Mdel V, Saavedra P, Quesada Gomez JM, Sosa Henriquez M. [High prevalence of hypovitaminosis D in medical students in Gran Canaria, Canary Islands (Spain)]. Endocrinol Nutr. 2011 Jun-Jul;58(6):267-73. doi: 10.1016/j.endonu.2011.03.002. Epub 2011 May 8. Spanish. PMID 21555257